CLINICAL TRIAL: NCT02696161
Title: The Long-term Effect of Platelet Rich Plasma and Perineural Injection Therapy in Patients With Carpal Tunnel Syndrome
Brief Title: Platelet Rich Plasma and Perineural Injection Therapy for Carpal Tunnel Syndrome
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Tri-Service General Hospital (Other)
Responsible Party: Principal Investigator, Yung-Tsan Wu, Attending Physician of Department of Physical Medicine and Rehabilitation, Tri-Service General Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: PRP for CTS
Record Dates: First submitted 2016-02-22; First posted 2016-03-02 (Estimated); Last update posted 2019-06-19 (Actual); Status verified 2019-06

CONDITIONS: Carpal Tunnel Syndrome
Keywords: platelet rich plasma; Perineural injection therapy
MeSH Terms: conditions — Carpal Tunnel Syndrome | interventions — Glucose

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- platelet rich plasma injection (Experimental): The platelet rich plasma (PRP) is a new and potential treatment for peripheral neuropathy in many animal studies.
  Interventions: Other: platelet rich plasma
- 5% dextrose (Placebo Comparator): 5% dextrose for hydrodissection
  Interventions: Other: 5% dextrose

INTERVENTIONS:
Other: platelet rich plasma — Ultrasound-guided 3cc PRP injection between proximal carpal tunnel and median nerve.
  Arms: platelet rich plasma injection
Other: 5% dextrose — Ultrasound-guided 3cc 5% dextrose injection between proximal carpal tunnel and median nerve.
  Arms: 5% dextrose

SUMMARY:
Carpal tunnel syndrome (CTS) is the most common peripheral entrapment neuropathy with involving compression of the median nerve in the carpal tunnel. Rather than other progressive disease, CTS is characterized by remission and recurrence. Although many conservative managements of CTS, the effectiveness of these methods is insignificant or only persist for a short duration. The platelet rich plasma (PRP) is a new and potential treatment for patients with kinds of musculoskeletal disorders and recent reports showed being beneficial for peripheral neuropathy in animal studies. Since 2014, two small clinical trials showed the positive effect of PRP in peripheral neuropathy. One study shown the PRP has therapeutic effect for peripheral neuropathy in patients with leprosy. In addition, PRP having protective effect against neurological deficit of facial nerve during superficial parotidectomy. However, these studies have not entirely proved the effects of PRP on peripheral neuropathy because these studies enrolled small number of patients and lacked controlled design. In addition, the PRP was not used for treating CTS so far. The investigators design a randomized, double-blind, controlled trail to assess the effect after ultrasound-guided PRP injection in patients with CTS.

DETAILED DESCRIPTION:
After obtaining written informed consent, patients of clinically diagnosed with CTS were randomized into intervention and control group. Participants in intervention group received one-dose ultrasound-guided PRP injection and control group received one-dose ultrasound-guided 5% dextrose injection. No additional treatment after injection through the study period. The primary outcome is visual analog scale (VAS) and secondary outcomes include Boston Carpal Tunnel Syndrome Questionnaire (BCTQ), cross-sectional area (CSA) of the median nerve, sensory nerve conduction velocity of the median nerve, and finger pinch strength. The evaluation was performed pretreatment as well as on the 2nd, 4th, 8th, 12th, 16th and 24th week after the treatment.

ELIGIBILITY:
Inclusion Criteria:

* Age between 20-80 year-old.
* Diagnosis was confirmed using an electrophysiological study

Exclusion Criteria:

* Cancer
* Coagulopathy
* Pregnancy
* Inflammation status
* Cervical radiculopathy
* Polyneuropathy, brachial plexopathy
* Thoracic outlet syndrome
* Previously undergone wrist surgery or steroid injection for CTS

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 52 (Actual)
Dates: Start 2016-02-01 (Actual); Primary Completion 2017-07-31 (Actual); Study Completion 2017-07-31 (Actual)

PRIMARY OUTCOMES:
Change from baseline in severity of symptoms and functional status on 2nd, 4th, 8th, 12th, 16th and 24th weeks after treatment. | Pre-treatment, 2nd, 4th, 8th, 12th, 16th and 24th weeks after treatment.
  Boston carpal tunnel syndrome questionnaire (BCTQ) is a frequently used patient-based questionnaire for measurement of CTS which encompasses two components. In total, 11 questions and 8 items were evaluated to rate the symptom severity scale (SSS) and functional status scale (FSS), respectively. Both subscales range from 1 to 5 with a higher score indicating a higher degree of disability. The mean of total SSS and FSS divided with each item score were used for further analysis.

SECONDARY OUTCOMES:
Change from baseline in cross-sectional area of the median nerve on 2nd, 4th, 8th, 12th, 16th and 24th weeks after treatment. | Pre-treatment, 2nd, 4th, 8th, 12th, 16th and 24th weeks after treatment.
  Using the musculoskeletal sonogram to measure the cross-sectional area of the median nerve.
Change from baseline in conduction velocity, amplitude of median nerve on 2nd, 4th, 8th, 12th, 16th and 24th weeks after treatment. | Pre-treatment, 2nd, 4th, 8th, 12th, 16th and 24th weeks after treatment.
  The antidromic sensory nerve conduction velocity of the median nerve was performed on all subjects according to the protocol reported by the American Academy of Neurology (USA). The median nerve was stimulated at the wrist between the palmar longus and flexor carpal radialis tendon at a distance of approximately 14 cm from the active electrode.
Change from baseline in finger pinch on 2nd, 4th, 8th, 12th, 16th and 24th weeks after treatment. | Pre-treatment, 2nd, 4th, 8th, 12th, 16th and 24th weeks after treatment.
  The finger pinch strength was measured using dynamometer (Fabrication Enterprises Inc., USA). The subject was seated with shoulder adducted and neutrally rotated with the elbow flexed at 90°. The forearm and wrist were positioned in a neutral position for the palmar pinch

CONTACTS AND LOCATIONS:
Overall Officials: Yung-Tsan Wu, MD., Principal Investigator — Department of Physical Medicine and Rehabilitation, Tri-Service General Hospital
Locations (1):
- Department of Physical Medicine and Rehabilitation, Tri-Service General Hospital, Taipei, Neihu District, Taiwan

IPD SHARING:
Plan to Share IPD: Yes

REFERENCES:
- [Result] Kucuk L, Gunay H, Erbas O, Kucuk U, Atamaz F, Coskunol E. Effects of platelet-rich plasma on nerve regeneration in a rat model. Acta Orthop Traumatol Turc. 2014;48(4):449-54. doi: 10.3944/AOTT.2014.13.0029. PMID 25230270
- [Result] Zheng C, Zhu Q, Liu X, Huang X, He C, Jiang L, Quan D, Zhou X, Zhu Z. Effect of platelet-rich plasma (PRP) concentration on proliferation, neurotrophic function and migration of Schwann cells in vitro. J Tissue Eng Regen Med. 2016 May;10(5):428-36. doi: 10.1002/term.1756. Epub 2013 May 31. PMID 23723151
- [Result] Lichtenfels M, Colome L, Sebben AD, Braga-Silva J. Effect of Platelet Rich Plasma and Platelet Rich Fibrin on sciatic nerve regeneration in a rat model. Microsurgery. 2013 Jul;33(5):383-90. doi: 10.1002/micr.22105. Epub 2013 May 2. PMID 23640879
- [Result] Park GY, Kwon DR. Platelet-rich plasma limits the nerve injury caused by 10% dextrose in the rabbit median nerve. Muscle Nerve. 2014 Jan;49(1):56-60. doi: 10.1002/mus.23863. Epub 2013 Sep 20. PMID 23558771
- [Result] Anjayani S, Wirohadidjojo YW, Adam AM, Suwandi D, Seweng A, Amiruddin MD. Sensory improvement of leprosy peripheral neuropathy in patients treated with perineural injection of platelet-rich plasma. Int J Dermatol. 2014 Jan;53(1):109-13. doi: 10.1111/ijd.12162. Epub 2013 Oct 29. PMID 24168291